CLINICAL TRIAL: NCT03997136
Title: Prognostic Impact of Surgical Resection Extent for Supratentorial High Grade Gliomas.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amr Badary, Resident Doctor, Assiut University
Other Study IDs: Brain Gliomas Surgery
Record Dates: First submitted 2019-06-21; First posted 2019-06-25 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Supratentorial Glioblastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Supratentorial high grade gliomas resection. — Total, near total or subtotal/debulking resection of the brain supratentorial high grade gliomas

SUMMARY:
Prospective randomized controlled clinical trials (single arm study) of surgical treatment modalities for supratentorial high grade gliomas within the next two years.

DETAILED DESCRIPTION:
Supratentorial high grade gliomas are for surgical resection in any case according to many factors.

Investigators will compare the outcomes/survival rate and clinical outcome of the different resection types (Total, near total, subtotal/debulking) of supratentorial high grade gliomas according to the clinical condition and comorbidities of the patient, the location and morphology of the lesion, the grading of lesions, and the clinical experience of the neurosurgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo surgical excision of the supratentorial high grade gliomas at the time of study (two years).
* Denovo disease for the first time.
* Any age

Exclusion Criteria:

* Low-grade Gliomas.
* Infratentorial high-grade gliomas.
* Past history of gliomas.
* Patients who are unfit for any neurosurgical interventions.
* Patients who do not receive their adjuvant standard therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases of patients of supratentorial high grade gliomas that fullfill the selection criteria that will be admitted in the department of neurosurgery in Assuit university hospital. (Non propability sample size) with expected size of 28 patients starting from 01/07/2019 to 15/06/2021.
  Patients whose follow-ups will be lost due to any other cause will be excluded from this study (expected to be 25%). Additionally, the competence of follow-up will be approved by imaging and medical records.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2019-09-01 (Estimated); Primary Completion 2021-04-01 (Estimated); Study Completion 2021-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical picture using Modified Rankin's Scale (mRS). | 1 year
  The changes in clinical condition of the patients will be assessed using Modified Rankin's Scale (mRS) before and after treatment.
  The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.

SECONDARY OUTCOMES:
Recurrence or increased residual | within 3 months after treatment
  Recurrence of the tumor

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Ragab, Study Director — Assiut University

REFERENCES:
- [Background] Gulati S, Jakola AS, Nerland US, Weber C, Solheim O. The risk of getting worse: surgically acquired deficits, perioperative complications, and functional outcomes after primary resection of glioblastoma. World Neurosurg. 2011 Dec;76(6):572-9. doi: 10.1016/j.wneu.2011.06.014. PMID 22251506
- [Background] Ostrom QT, Bauchet L, Davis FG, Deltour I, Fisher JL, Langer CE, Pekmezci M, Schwartzbaum JA, Turner MC, Walsh KM, Wrensch MR, Barnholtz-Sloan JS. The epidemiology of glioma in adults: a "state of the science" review. Neuro Oncol. 2014 Jul;16(7):896-913. doi: 10.1093/neuonc/nou087. PMID 24842956
- [Background] Ryken TC, Frankel B, Julien T, Olson JJ. Surgical management of newly diagnosed glioblastoma in adults: role of cytoreductive surgery. J Neurooncol. 2008 Sep;89(3):271-86. doi: 10.1007/s11060-008-9614-5. Epub 2008 Aug 20. No abstract available. PMID 18712281
- [Background] Sanai N, Polley MY, McDermott MW, Parsa AT, Berger MS. An extent of resection threshold for newly diagnosed glioblastomas. J Neurosurg. 2011 Jul;115(1):3-8. doi: 10.3171/2011.2.jns10998. Epub 2011 Mar 18. PMID 21417701
- [Background] Orringer D, Lau D, Khatri S, Zamora-Berridi GJ, Zhang K, Wu C, Chaudhary N, Sagher O. Extent of resection in patients with glioblastoma: limiting factors, perception of resectability, and effect on survival. J Neurosurg. 2012 Nov;117(5):851-9. doi: 10.3171/2012.8.JNS12234. Epub 2012 Sep 14. PMID 22978537